CLINICAL TRIAL: NCT06081426
Title: Elucidating Neurobiological Mechanisms Underlying the Therapeutic Effect of the Ketogenic Diet in Bipolar Disorder (BD): a Multidisciplinary Mechanistic Study
Brief Title: Examining Neurobiological Mechanisms Underlying the Therapeutic Effect of the Ketogenic Diet in Bipolar Disorder (BD)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Collaborators: Baszucki Brain Research Fund (Other)
Responsible Party: Principal Investigator, Mary Phillips, MD MD (Cantab), Professor, University of Pittsburgh
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: STUDY23080048
Record Dates: First submitted 2023-09-22; First posted 2023-10-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Bipolar Disorder
Keywords: Ketogenic Diet; Magnetic Resonance Imaging
MeSH Terms: conditions — Bipolar Disorder | interventions — Diet, Ketogenic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1st phase Non-ketogenic Diet / 2nd phase Ketogenic Diet (Experimental): Participants with Bipolar Disorder will consume a non-ketogenic diet for the first phase of the study and then a ketogenic diet for the second phase of the study
  Interventions: Other: Non-ketogenic Diet; Other: Ketogenic Diet
- 1st phase Ketogenic Diet / 2nd phase Non-ketogenic Diet (Experimental): Participants with Bipolar Disorder will consume a ketogenic diet for the first phase of the study and then a non-ketogenic diet for the second phase of the study
  Interventions: Other: Non-ketogenic Diet; Other: Ketogenic Diet
- No diet (Other): Participants without Bipolar Disorder will not participate in the diet phases of the study
  Interventions: Other: No diet

INTERVENTIONS:
Other: Non-ketogenic Diet — Consuming a non-ketogenic diet
  Arms: 1st phase Ketogenic Diet / 2nd phase Non-ketogenic Diet; 1st phase Non-ketogenic Diet / 2nd phase Ketogenic Diet
Other: Ketogenic Diet — Consuming a ketogenic diet
  Arms: 1st phase Ketogenic Diet / 2nd phase Non-ketogenic Diet; 1st phase Non-ketogenic Diet / 2nd phase Ketogenic Diet
Other: No diet — Participants without Bipolar Disorder will not participate in the diet phases of the study
  Arms: No diet

SUMMARY:
The investigators aim to examine the effect of the ketogenic diet on brain activity, metabolism, and emotions in adults with Bipolar Disorder (BD).

DETAILED DESCRIPTION:
The investigators hypothesize that a ketogenic diet will enhance levels of the ketone body β-Hydroxybutyrate (beta OHB), resulting in reduced mania/hypomania severity and predisposition to mania/hypomania in individuals with BD. To test this hypothesis in depth, the investigators will use a novel, multidisciplinary mechanistic study using multimodal neuroimaging, peripheral markers of mitochondrial metabolism, and participant-derived induced pluripotent stem cell (iPSC)-derived organoids.

ELIGIBILITY:
Inclusion Criteria:

All participants:

* 18-40 years of age
* Not following a ketogenic diet

BD hypomanic group (n=30):

* Meeting sex proportion: 50% female
* Meeting diagnosis proportion: 50:50% Bipolar I: Bipolar II (BDI:II) (Diagnostic and Statistical Manual of Mental Disorders 5; DSM-5)
* Score greater than 10 on the Young Mania Rating Scale score(YMRS)
* BD medications will be allowed as in our previous studies: any combination of atypical antipsychotics, lithium, antidepressants, anxiolytics (common in BD)

BD euthymic group (n=30):

* Meeting sex proportion: 50% female
* Meeting diagnosis proportion: 50:50% BDI:II (DSM-5)
* Score less than or equal to 10 on YMRS
* BD medications will be allowed as in our previous studies: any combination of atypical antipsychotics, lithium, antidepressants, anxiolytics (common in BD)

Healthy Control (HC) Group (n=30):

* Sex matched with BD groups
* No psychiatric history

Exclusion Criteria:

All participants:

* Not between 18-40 years of age
* History of head injury, neurological, pervasive developmental disorder (e.g. autism), systemic medical disease and treatment (medical records, participant report)
* Mini-Mental State Examination score (cognitive state) <24
* Premorbid National Adult Reading Test Intelligent Quotient (NAART IQ) estimate<85
* Visual disturbance: <20/40 Snellen visual acuity
* History of alcohol/substance use disorder (SUD; all substances, including nicotine), and/or illicit substance use (except cannabis) over the last 6 months (SCID-5). Note: lifetime/present cannabis use (at non-abuse (<3 times in the past month) and non SUD levels) will be allowed, given its common usage in BD and young adults. Cannabis SUD over the last 6 months will not be allowed. Urine tests on scan days will exclude current illicit substance use (except cannabis). Salivary alcohol tests on scan days will exclude intoxicated individuals
* MRI exclusion: metallic objects, e.g., surgical implants; claustrophobia; positive pregnancy test for females or self-report pregnancy
* Unable to understand English
* Conditions related to the pancreas, liver, thyroid or gallbladder.
* Taking anticoagulants and/or those with blood dyscrasias (illnesses) who have coagulation disorders (eg, hemophilia) because of the ketomojo finger stick blood tests
* Scoring 3 or higher on positive symptom factor questions on the Positive and Negative Syndrome Scale (PANSS) questionnaire (indicative of psychotic symptoms)
* Currently following a ketogenic diet
* Head circumference larger than 24 inches (62cm) and/or chest circumference larger than 55 inches (139 cm)

BD hypomanic group:

* Must be meeting sex proportions: not 50% female
* Must be meeting diagnosis proportions: not 50:50% BDI:II (DSM-5)
* Diagnosis of BD in a manic or euthymic episode
* Score 10 or lower on the Young Mania Rating Scale score(YMRS)
* Using psychotropic medications other than those allowed in inclusion criteria
* Does not have a smartphone with a) iOS version 12.0 or above, or b) Android version 8 and later to use with the Keto-Mojo app

BD euthymic group:

* Not meeting sex proportion: not 50% female
* Not meeting diagnosis proportion: not 50:50% BDI:II
* Diagnosis of BD in a depressive, hypomanic, or manic episode
* Score greater than 10 on YMRS
* Using psychotropic medications other than those allowed in inclusion criteria
* Does not have a smartphone with a) iOS version 12.0 or above, or b) Android version 8 and later to use with the Keto-Mojo app

Healthy Control (HC) Group

* Not sex-matched with BD groups
* Has psychiatric history

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 107 (Estimated)
Dates: Start 2024-01-12 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Blood oxygen level-dependent (BOLD) signal at Scan 1 | Baseline Scan 1 (all participants)
  The blood oxygen level-dependent (BOLD) signal indicates brain activity and connectivity
Blood oxygen level-dependent (BOLD) signal at Scan 2 | End of first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  The blood oxygen level-dependent (BOLD) signal indicates brain activity and connectivity
Blood oxygen level-dependent (BOLD) signal at Scan 3 | End of second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  The blood oxygen level-dependent (BOLD) signal indicates brain activity and connectivity
Manic symptoms at Scan 1 | Baseline Scan 1 (all participants)
  The Young Mania Rating Scale (YMRS) indicates the level of manic symptoms with a total score that varies between zero (better outcome) and 60 (worse outcome)
Manic symptoms at Scan 2 | Scan 2 at end of first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  The Young Mania Rating Scale (YMRS) indicates the level of manic symptoms with a total score that varies between zero (better outcome) and 60 (worse outcome)
Manic symptoms at Scan 3 | Scan 3 at end of second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  The Young Mania Rating Scale (YMRS) indicates the level of manic symptoms with a total score that varies between zero (better outcome) and 60 (worse outcome)
Fasting Glucose at Baseline | Baseline (all participants)
  Fasting glucose blood levels
Fasting lipids at Baseline | Baseline (all participants)
  Fasting lipid blood levels
Fasting hepatic function panel at Baseline: total protein | Baseline (all participants)
  Fasting levels of total protein in the blood
Fasting hepatic function panel at Baseline: albumin | Baseline (all participants)
  Fasting levels of albumin in the blood
Fasting hepatic function panel at Baseline: bilirubin | Baseline (all participants)
  Fasting levels of bilirubin in the blood
Fasting hepatic function panel at Baseline: liver enzyme | Baseline (all participants)
  Fasting levels of liver enzyme in the blood
Fasting Glucose at halfway point through first dietary phase | Halfway point through first dietary phase (4-5 weeks) (participants with Bipolar Disorder)
  Fasting glucose blood levels
Fasting lipids at halfway point through first dietary phase | Halfway point through first dietary phase (4-5 weeks) (participants with Bipolar Disorder)
  Fasting lipid blood levels
Fasting hepatic function at halfway point through first dietary phase: total protein | Halfway point through first dietary phase (4-5 weeks) (participants with Bipolar Disorder)
  Fasting levels of total protein in the blood
Fasting hepatic function at halfway point through first dietary phase: albumin | Halfway point through first dietary phase (4-5 weeks) (participants with Bipolar Disorder)
  Fasting levels of albumin in the blood
Fasting hepatic function at halfway point through first dietary phase: bilirubin | Halfway point through first dietary phase (4-5 weeks) (participants with Bipolar Disorder)
  Fasting levels of bilirubin in the blood
Fasting hepatic function at halfway point through first dietary phase: liver enzyme | Halfway point through first dietary phase (4-5 weeks) (participants with Bipolar Disorder)
  Fasting levels of liver enzyme in the blood
Fasting Glucose at end of first dietary phase | End of first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Fasting glucose blood levels
Fasting lipids at end of first dietary phase | End of first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Fasting lipid blood levels
Fasting hepatic function at end of first dietary phase: total protein | End of first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Fasting levels of total protein in the blood
Fasting hepatic function at end of first dietary phase: albumin | End of first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Fasting levels of albumin in the blood
Fasting hepatic function at end of first dietary phase: bilirubin | End of first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Fasting levels of bilirubin in the blood
Fasting hepatic function at end of first dietary phase: liver enzyme | End of first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Fasting levels of liver enzyme in the blood
Fasting Glucose at halfway point through second dietary phase | Halfway point through second dietary phase (4-5 weeks) (participants with Bipolar Disorder)
  Fasting glucose blood levels
Fasting lipids at halfway point through second dietary phase | Halfway point through second dietary phase (4-5 weeks) (participants with Bipolar Disorder)
  Fasting lipid blood levels
Fasting hepatic function at halfway point through second dietary phase: total protein | Halfway point through second dietary phase (4-5 weeks) (participants with Bipolar Disorder)
  Fasting levels of total protein in the blood
Fasting hepatic function at halfway point through second dietary phase: albumin | Halfway point through second dietary phase (4-5 weeks) (participants with Bipolar Disorder)
  Fasting levels of albumin in the blood
Fasting hepatic function at halfway point through second dietary phase: bilirubin | Halfway point through second dietary phase (4-5 weeks) (participants with Bipolar Disorder)
  Fasting levels of bilirubin in the blood
Fasting hepatic function at halfway point through second dietary phase: liver enzyme | Halfway point through second dietary phase (4-5 weeks) (participants with Bipolar Disorder)
  Fasting levels of liver enzyme in the blood
Fasting Glucose at end of second dietary phase | End of second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Fasting glucose blood levels
Fasting lipids at end of second dietary phase | End of second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Fasting lipids blood levels
Fasting hepatic function at end of second dietary phase: total protein | End of second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Fasting levels of total protein in the blood
Fasting hepatic function at end of second dietary phase: albumin | End of second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Fasting levels of albumin in the blood
Fasting hepatic function at end of second dietary phase: bilirubin | End of second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Fasting levels of bilirubin in the blood
Fasting hepatic function at end of second dietary phase: liver enzyme | End of second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Fasting levels of liver enzyme in the blood
Gamma-aminobutyric acid (GABA) at Baseline | Baseline Scan 1 (all participants)
  Gamma-aminobutyric acid (GABA) concentrations in the brain
Glutamate at Baseline | Baseline Scan 1 (all participants)
  Glutamate concentrations in the brain
Lactate at Baseline | Baseline Scan 1 (all participants)
  Lactate concentrations in the brain
Gamma-aminobutyric acid (GABA) at end of first dietary phase | Scan 2 at end of first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Gamma-aminobutyric acid (GABA) concentrations in the brain
Glutamate at end of first dietary phase | Scan 2 at end of first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Glutamate concentrations in the brain
Lactate at end of first dietary phase | Scan 2 at end of first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Lactate concentrations in the brain
Gamma-aminobutyric acid (GABA) at end of second dietary phase | Scan 3 at end of second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Gamma-aminobutyric acid (GABA) concentrations in the brain
Glutamate at end of second dietary phase | Scan 3 at end of second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Glutamate concentrations in the brain
Lactate at end of second dietary phase | Scan 3 at end of second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Lactate concentrations in the brain

SECONDARY OUTCOMES:
Average total sleep time during Ketogenic vs Normal diet | Wrist actigraphy will be collected throughout the 8-10wk ketogenic diet and normal diet study intervals
  Total sleep time will be assessed using wrist actigraphy. Wrist actigraphy will be collected continuously, at-home.
Average rest-activity rhythm interdaily stability during Ketogenic vs Normal diet | Wrist actigraphy will be collected throughout the 8-10 wk ketogenic diet and normal diet study intervals.
  Rest-activity rhythm interdaily stability will be assessed using wrist actigraphy. Wrist actigraphy will be collected continuously, at-home
Ecological momentary assessments (EMA) during the first dietary phase: Mood monitoring | The first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Mood monitoring in real time in participants with Bipolar Disorder: rate mood on a scale of 1-7 with 1 being very low mood and 7 being very high mood
Ecological momentary assessments (EMA) during the first dietary phase: Energy monitoring | The first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Energy monitoring in real time in participants with Bipolar Disorder: rate energy on a scale of 1-7 with 1 being very low energy and 7 being very high energy
Ecological momentary assessments (EMA) during the first dietary phase: Suicidality monitoring | The first dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Suicidality monitoring in real time in participants with Bipolar Disorder: answer yes or no to having self-harm/suicide thoughts and plans
Ecological momentary assessments (EMA) during the second dietary phase: Mood monitoring | The second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Mood monitoring in real time in participants with Bipolar Disorder: rate mood on a scale of 1-7 with 1 being very low mood and 7 being very high mood
Ecological momentary assessments (EMA) during the second dietary phase: Energy monitoring | The second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Energy monitoring in real time in participants with Bipolar Disorder: rate energy on a scale of 1-7 with 1 being very low energy and 7 being very high energy
Ecological momentary assessments (EMA) during the second dietary phase: Suicidality monitoring | The second dietary phase (8-10 weeks) (participants with Bipolar Disorder)
  Suicidality monitoring in real time in participants with Bipolar Disorder: answer yes or no to having self-harm/suicide thoughts and plans

CONTACTS AND LOCATIONS:
Overall Officials: Mary Phillips, MD, Principal Investigator — University of Pittsburgh
Locations (1):
- University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Yes
Informed consent will be collected from study participants that allows for broad sharing of participants' de-identified data. Data transfer procedures will be in accordance with all Institutional Review Board guidelines and federal regulations including HIPAA (Health Insurance Portability and Accountability Act of 1996).
Time Frame: The principal investigators (PIs) reserve the right to publish on the stated aims in a timely manner. Data will be available for addressing other research questions (i.e. which are not described in funded/pending grants) as soon as the data have been checked for accuracy (a period which will be no later than one year after the completion of each assessment). After the study has ended, the study investigators will continue to test the stated aims, but will also continue to solicit collaborations with outside researchers and to consider data requests in a timely manner.
Access Criteria: Outside investigators must submit a 1)proposal of the study aims, hypotheses, variables/constructs, analytic approach, and estimated duration of the proposed research; 2)resume, qualifications, source of financial support, and conflict of interest statement; 3)sign a data-sharing agreement and confidentiality statement that stipulates using the data for the stated research purposes only, securing the data using appropriate computer technology, not manipulating the data in order to identify participants, acknowledging the grant that supported data collection and management in publications/presentations, and destroying or returning the data after analyses are complete; 4)obtain approval from their Institutional Review Board, and along with other staff members who have access to the data, submit certificates of the University of Pittsburgh Education and Certification Program in Research Practice Fundamentals or provide written documentation of similar human subjects protection training.